CLINICAL TRIAL: NCT00737217
Title: Executive, Activities of Daily Living, and Cholinergic Functions in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Nicolaas Bohnen, MD, PhD, Principal Investigator, University of Michigan
Other Study IDs: 2005-0464
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's disease
  Interventions: Behavioral: Behavioral assessment/questionnaire
- Normal Controls
  Interventions: Behavioral: Behavioral assessment/questionnaire

INTERVENTIONS:
Behavioral: Behavioral assessment/questionnaire — Complete behavioral assessment/questionnaire

SUMMARY:
This research study will evaluate functions of memory, thinking, behavior, and daily life activities and how these relate to the measurement of certain chemicals (acetylcholine and dopamine) in the brain using an imaging procedure called positron emission tomography (PET). You may know that in Alzheimer's dementia (dementia is a disease where persons become forgetful and confused), a reduction in the amount of acetylcholine, a "neurotransmitter" substance (a chemical messenger that nerve cells need to communicate with each other), may be responsible for some of the memory and behavioral changes. At the present time, the investigators have no clear information on the levels of acetylcholine in the brain of patients with Parkinson's disease who also have memory or behavioral changes.

ELIGIBILITY:
Inclusion Criteria:

* PDD: Patients who meet the UK Parkinson's Disease Society Brain Bank Research Center (UKPDSBRC) clinical diagnostic criteria for PD with dementia (MMSE 18-25; n=28; age 50-85 years; M/F) are eligible for the study. Hoehn and Yahr stages I-III.
* PD. Patients with who meet the UKPDSBRC criteria for PD with a MMSE of >25 (n=28; age 50-85 years; M/F). Hoehn and Yahr stages I-III.
* Normal control subjects (n=16) (age 50-85 years; M/F).
* No current or past history of neurologic or psychiatric illness.

Exclusion Criteria:

* Any subjects on cholinergic, anti-cholinergic drugs will be excluded from the study.
* Current or past history of neurologic or psychiatric illness.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease, either with or without memory or concentration difficulties, and normal control persons between the ages of 50-85 years are eligible to participate in this study. Participants should be willing and able to comply with study requirements. Normal control persons should not have a history of brain or mental disorders. Both males and females are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2006-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Functional, Cognitive and Mobility Laboratory, Ann Arbor, Michigan, United States